CLINICAL TRIAL: NCT06899464
Title: Safety and Feasibility of Using Cerebrolysin in the Treatment of Primary Intracerebral Hemorrhage
Brief Title: Safety and Feasibility of Using Cerebrolysin in the Treatment of Primary Intracerebral Hemorrhage - a Prospective Randomized Open Blinded End-point Trial
Acronym: CLINCH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cardinal Stefan Wyszynski University (Other)
Responsible Party: Principal Investigator, Adam Kobayashi, MD PhD, Cardinal Stefan Wyszynski University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000101
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Intracerebral Hemorrhage; Hemorrhagic Stroke, Intracerebral; Hemorrhagic Stroke; Stroke
Keywords: Cerebrolysin in stroke; neuroprotection in stroke; Cerebrolysin in hemorrhagic stroke
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhagic Stroke; Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerebrolysin (Experimental): Cerebrolysin infusion (50 ml mixed with 250 mL of saline) will be initiated as soon as possible and within 6 hours of stroke onset. Cerebrolysin treatment will be continued (50 ml/d) once daily until day 14.
  Interventions: Drug: 14-day Cerebrolysin treatment
- Placebo (Placebo Comparator): Standard of care
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Drug: 14-day Cerebrolysin treatment — 14-day cerebrolysin treatment initiated within 6 hours of onset of stroke
  Arms: Cerebrolysin
Other: Standard of Care (SOC) — Standard of care treatment
  Arms: Placebo

SUMMARY:
This study is designed to determine the safety and feasibility of using Cerebrolysin in treating primary intracerebral hemorrhage (ICH).

This is a multicenter, prospective, randomized, open-label, blinded end-point, phase IV parallel group study done in specialized stroke treatment centers in Poland. The study objective is to evaluate if a 14-day cerebrolysin treatment initiated within 6 hours of onset of primary lobar hemorrhage in addition to the standard of care that includes early intensive rehabilitation is safe and feasible, affects hematoma growth and improves the outcome.

This study is designed to assess the early effect of using Cerebrolysin in patients after ICH, therefore 3 months of follow-up has been chosen. Patients will receive 50 ml of Cerebrolysin once daily until day 14. Subjects will be evaluated on Day 1 (baseline), Day 2, Day 7, Day 30 and Day 90.

Enrollment to the study is expected to reach 30 subjects in 12 months. The study should be completed within 15 months (the end of study).

The primary outcome measure will be change from baseline in functional independence (mRS 0-2) at Day 90 following stroke onset. The safety outcome will be the number of serious adverse events until Day 30.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* NIHSS ≥8 at randomization
* Stroke onset <6h
* Pre-randomization head CT demonstrating an acute, primary lobar ICH
* ICH volume 30 to 80 mL
* Glasgow Coma Score (GCS) 5 to 12
* Pre-stroke independence (modified Rankin Score 0 to 2)
* Ability to provide informed consent
* No history of prior stroke

Exclusion Criteria:

* Hemorrhage caused by head trauma
* Medical history or neuroimaging findings suggestive of ruptured aneurysm, arteriovenous malformation (AVM), vascular anomaly, Moyamoya disease, venous sinus thrombosis, mass or tumor, hemorrhagic conversion of an ischemic infarct
* Bilateral fixed dilated pupils
* Extensor motor posturing
* Intraventricular extension of the hemorrhage is visually estimated to involve >50% of either of the lateral ventricles
* Primary Thalamic and basal ganglia ICH
* Infratentorial intraparenchymal hemorrhage including midbrain, pontine, or cerebellar
* Current use of low molecular weight heparins in therapeutic dose
* Evidence of active bleeding
* Uncorrected coagulopathy or known clotting disorder
* Platelet count < 75,000, International Normalized Ratio (INR) > 1.4 after correction
* End stage renal disease
* Patients with a mechanical heart valve
* End-stage liver disease
* Epilepsy with grand mal seizures
* History of drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Positive urine or serum pregnancy test in female subjects without documented history of surgical sterilization or post-menopausal
* Known life-expectancy of less than 6 months
* No reasonable expectation of recovery, Do-Not-Resuscitate (DNR), or comfort measures only prior to randomization
* Participation in a concurrent interventional medical investigation or clinical trial
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent
* Any condition that would represent a contraindication for cerebrolysin administration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy Outcome | 90 days from stroke onset
  Change from baseline in functional independence (mRS 0-2) at Day 90 following stroke onset
Safety Outcome | 30 days from stroke onset
  Number of Serious Adverse Events until Day 30

SECONDARY OUTCOMES:
Neurological deficit | Day 2, 7, 30, and 90 from stroke onset
  Change from baseline in neurological deficit measured by NIHSS at Day 2, 7, 30, and 90
Functional independence | 30 days from stroke onset
  Change from baseline in improving functional independence (mRS 0-2) at Day 30
Activities of daily living | 30 and 90 days from stroke onset
  Change from baseline in activities of daily living (by BartheI Index) on Day 30 and 90
Hematoma growth | 2 days from stroke onset
  Hematoma growth from Day 1 to Day 2
Mortality | 90 days from stroke onset
  Mortality rate on Day 90

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR